CLINICAL TRIAL: NCT01121744
Title: Supralimus-Core™ Pharmacokinetic (PK) Study: Evaluation of Pharmacokinetic (PK) and Safety of the Supralimus-Core™ Sirolimus Eluting Coronary Stent System in De Novo Native Coronary Artery Lesions
Brief Title: Supralimus-Core™ Pharmacokinetic (PK) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Responsible Party: Dr. Atul Abhyankar, Sahajanand Medical Technologies Pvt. Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC001:V.1.0:Dated 12/12/2008.
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Drug Eluting Stents (DES); Pharmacokinetic (PK)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Supralimus-Core™ Sirolimus eluting Coronary Stent — Supralimus-Core™ Coronary Stent System consisting of the Coronnium® coronary stent (CE approved) having Biodegradable Polymeric Matrix on a Co-Cr alloy Platform. Sirolimus Drug concentration is 1.4 µg/mm2.
  Other Names: Drug Eluting Stent (DES)

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetic (PK) and safety associated with Supralimus-Core™ Sirolimus Eluting Coronary Stent system in the treatment of single de novo lesions in native coronary arteries between 2.5 to 3.5 mm in diameter.

DETAILED DESCRIPTION:
This is a multi-centric, interventional, non-randomized, open label, Uncontrolled, single group assignment, Pharmacokinetics study. Approximately 20 patients will be enrolled in the study. Patients will be followed for 48 days post-procedure.

ELIGIBILITY:
Patients with de novo native coronary artery lesions located in epicardial vessel who qualify for percutaneous coronary intervention will be included according to the inclusion and exclusion criteria specified below:

Inclusion Criteria:

1. Age ≥18 years.
2. Eligible for percutaneous coronary intervention (PCI)
3. Acceptable candidate for CABG
4. Clinical evidence of ischemic heart disease and/or a positive territorial functional study. Documented stable angina pectoris ((Canadian Cardiovascular Society (CCS) Classification 1, 2, 3 or 4) or unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C or IIIB-C), or documented silent ischemia.
5. The target lesion is a single de novo coronary artery lesion with ≥ 50% and < 100% stenosis in one of the major epicardial territories (LAD, LCX or RCA). A second target lesion in another major epicardial vessel could be treated and this second lesion should fit with the inclusion/exclusion criteria and will receive the same type of stent.
6. The target lesion must be covered by one study stent, preferably with a margin of 3 mm on each side of the lesion.
7. The target lesion must be ≤ 34 mm in length by visual estimate.
8. The target reference vessel diameter must be ≥ 2.5 mm and ≤ 3.5 mm.
9. Patient or patient's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as notified / approved by the Institutional Review Board/Ethics Committee of the clinical site.

Exclusion Criteria:

1. Female of childbearing potential
2. Documented left ventricular ejection fraction (LVEF) ≤ 25%
3. Evidence of an acute Q-wave or non-Q-wave myocardial infarction within 72 hours preceding the index procedure
4. Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix®, Ceruvin) or ticlopidine (Ticlid®), heparin, sirolimus, cobalt chromium, contrast agent (that cannot be adequately pre-medicated)
5. A platelet count <100,000 cells/mm3 or >700,000 cells/mm3 or a WBC <3,000 cells/mm3
6. Acute or chronic renal dysfunction (creatinine >2.0mg/dl or >150µmol/L)
7. Target vessel has evidence of thrombus
8. Target vessel is excessively tortuous which makes it unsuitable for proper stent delivery and deployment
9. Previous bare metal stenting (less than 1 year) anywhere within the target vessel
10. Previous drug-eluting stenting anywhere within any epicardial vessel
11. The target lesion requires treatment with a device other than PTCA prior to stent placement (e.g. but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.)
12. Significant (>50%) stenosis proximal or distal to the target lesion that might require revascularization or impede run-off
13. Heavily calcified lesion and/or calcified lesion which cannot be successfully predilated
14. Target lesion is located in or supplied by an arterial or venous bypass graft
15. Ostial target lesion
16. Patient is currently participating in an investigational drug or device study, including its follow-up period
17. Within 30 days prior to procedure, patient has undergone a previous coronary interventional procedure of any kind
18. Within 48 days post-procedure, patient requires planned interventional treatment of any non-target vessel. Planned intervention of the target vessel after the index procedure is not allowed.
19. CVA within previous 6 months
20. Unprotected Left Main (LM) coronary artery disease (stenosis >50%)
21. In the investigator's opinion, patient has a co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
22. Planned surgery within 48 days after the index procedure
23. Life expectancy less than 1 year
24. Any contraindication to blood sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Cmax, Tmax, AUC24h, AUClast, AUC∞, λz, t½term, CL | Up to 48 days

SECONDARY OUTCOMES:
Major Adverse Cardiac Event (MACE) | Up to 48 days

CONTACTS AND LOCATIONS:
Locations (4):
- India (4):
  - Life Care Institute of Medical Science & research, Ahmedabad, Gujarat
  - Shree B. D. Mahavir Heart Institute, Surat, Gujarat
  - Baroda Heart Institute & Research Center, Vadodara, Gujarat
  - Bankers Heart Institute, Vadodara, Gujarat

REFERENCES:
- [Result] Thakkar AS, Abhyankar AD, Dani SI, Banker DN, Singh PI, Parmar SA, Mehta AA. Systemic exposure of sirolimus after coronary stent implantation in patients with de novo coronary lesions: Supralimus-Core(R) pharmacokinetic study. Indian Heart J. 2012 May-Jun;64(3):273-9. doi: 10.1016/S0019-4832(12)60086-8. PMID 22664810